CLINICAL TRIAL: NCT04136652
Title: Vaginal CO2 Laser for Stress Incontinence: A Randomized Controlled Trial
Brief Title: Vaginal CO2 Laser for Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Hrefna Bóel Sigurdardóttir, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-19013894
Record Dates: First submitted 2019-10-10; First posted 2019-10-23 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Stress Incontinence Female; Laser
Keywords: vaginal laser CO2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Only the doctor who performs the laser procedure knows which treatment the participant gets. The data analyzer will also know, in data analyses after all treatments are done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Placebo Comparator): The women are randomized, by a computer program, to a sham laser-treatment with the laser not active.
  Interventions: Procedure: CO2 laser- treatment (DEKA SmartXide2 Laser System, MonaLisa Touch
- Laser (Active Comparator): The women are randomized, by a computer program, to a vaginal CO2 laser-treatment with 30 w.
  Interventions: Procedure: CO2 laser- treatment (DEKA SmartXide2 Laser System, MonaLisa Touch

INTERVENTIONS:
Procedure: CO2 laser- treatment (DEKA SmartXide2 Laser System, MonaLisa Touch — women will receive a series of three treatments using a fractional (pulsed) CO2 laser system (SmartXide2 MonaLisa Touch, DEKA M.E.L.A Srl, Florence, Italy), each performed in an outpatient setting without analgesia. A tubular laser-probe is inserted in the vaginal canal until reaching the vaginal vault. A burst of laser pulses is transmitted through the probe and deflected at 90degrees in four directions towards the vaginal wall, then rotated 45degree for a second burst of pulses. Guided by markings on the probe, it is withdrawn 4mm and the procedure is repeated until reaching the introitus. Treatment parameters include power 30W, dwell time 1000us, 1000um spacing, using normal scan mode, with Smartstack setting for 1 at first application and 3 for the next two applications.

SUMMARY:
Our aim with this study is to determine if transvaginal CO2 laser- treatment (DEKA SmartXide2 Laser System, MonaLisa Touch), renders significant effect in women with SUI. To best test this hypothesis, the study will be performed in a prospective, randomised controlled fashion in our institution. We will measure the effect as patient reported improvement using a validated scale (ICIQ-UI SF) as well as an objective measurement (stress test)

DETAILED DESCRIPTION:
Patient will be included from our hospital (a Danish academic hospital) among women referred with incontinence. Eligible patients will be randomized to either laser treatment or "sham" laser treatment.

The study will take place in the department of Gynecology and Obstetrics of Hvidovre University Hospital, Copenhagen Denmark in the period of October 2019 to October 2020. Inclusion criteria for the study cohort and controls will be patients, referred from specialist gynecologists or GPs with SUI, that speak and understand Danish, are found without clinical relevant urogenital prolapse (grad 2 at maximum in al compartments), older than 18 years of age, with BMI under 35 and present with mild to moderate SUI evaluated after ICIQ-UI-SF (slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21). Exclusion criteria presence of pelvic organ prolapse greater than stage II, previous pelvic surgery for incontinence or prolaps, current infections, keloid formation, vaginal pain, dyspareunia, ICIQ-UI-SF>=19 (very severe) and ongoing pregnancy.

In this study, women will receive a series of three treatments using a fractional (pulsed) CO2 laser system (SmartXide2 MonaLisa Touch, DEKA M.E.L.A Srl, Florence, Italy), each performed in an outpatient setting without analgesia. A tubular laser-probe is inserted in the vaginal canal until reaching the vaginal vault. A burst of laser pulses is transmitted through the probe and deflected at 90degree in four directions towards the vaginal wall, then rotated 45 degrees for a second burst of pulses. Guided by markings on the probe, it is withdrawn 4mm and the procedure is repeated until reaching the introitus. Treatment parameters include power 30W, dwell time 1000us, 1000um spacing, using normal scan mode, with Smartstack setting for 1 at first application and 3 for the next two applications.

Both study- and placebo- treatments will be performed by specialist gynecologists employed in the department. Patients, who meet inclusion criteria and consent to study participation, will be randomized by computer service to conservative treatment, which encompass local estrogens (Vagifem 10ug twice weekly) if relevant (postmenopausal women) and pelvic floor training supervised by specialised physiotherapists in our own institution, whilst the study cohort will receive the same treatment with the addition of transvaginal laser applied thrice with 25- 45 days apart (CO2 laser- treatment (DEKA SmartXide2 Laser System, MonaLisa Touch). The controls will receive placebo treatment, with the use of the inactive laser, but relevant sound effects.

Primary outcome of the study is patient experienced improvement of SUI evaluated by standardized ICIQ-UI-SF questionnaire.

Our secondary outcome is objective improvement as measured by standardized stress test performed by specialist nurse before treatment and 1-2 month after last laser or placebo treatment. The bladder is emptied with a catheter and 300ml of saline is inserted. The patient is then stood up wearing a pad with legs slightly apart and asked to forcefully cough 10 timers, jump 10 times and make 10 squats. The examiner registers whether there is incontinence as either yes or no as well as grams of urin leakage in the pad. Furthermore, side- effects both positive and negative as well as patient satisfaction will be registered by the use of patient questionnaires at 1-2 months post treatment.

ELIGIBILITY:
Inclusion criteria

* referred from specialist gynecologists or GPs with SUI
* speak and understand Danish
* are found without clinical relevant urogenital prolapse
* older than 18 years of age
* with BMI under 35
* Present with mild to moderate SUI evaluated after ICIQ-UI-SF (slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21))

Exclusion criteria

* presence of pelvic organ prolapse greater than stage II
* previous pelvic surgery for prolapse or incontinence,
* current infections,
* keloid formation
* vaginal pain
* dyspareunia,
* ICIQ-UI-SF>=19 (very severe)
* ongoing pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
ICIQ-UI SF | Through study completion, an average of 6-8 months
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. Women will answer this questionnaire before they are booked for the first laser treatment. After al three treatments, they will have a control visit in an outpatient setting, where they fill out the questionaire again.

SECONDARY OUTCOMES:
Standardized stress test | Through study completion, an average of 6-8 months
  Objective improvement as measured by standardized stress test performed by specialist nurse before treatment and 1-2 month after last laser or placebo treatment. The bladder is emptied with a catheter and 300ml of saline is inserted. The patient is then stood up wearing a pad with legs slightly apart and asked to forcefully cough 10 times, jump 10 times and do 10 squats. The examiner registers whether there is incontinence as either yes or no as well as grams of urin leakage in the pad

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe B Schroll, MD, PhD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sigurdardottir HB, Kirschner B, Obel J, Aziz M, Stenz CB, Schroll JB. Vaginal CO2 laser treatment for urinary stress incontinence: A randomized controlled trial. Maturitas. 2025 Aug;199:108658. doi: 10.1016/j.maturitas.2025.108658. Epub 2025 Jul 3. PMID 40617073

DOCUMENTS (1):
  • Study Protocol (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT04136652/Prot_000.pdf